CLINICAL TRIAL: NCT02352584
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Parallel Phase III Study to Investigate the Efficacy(Immunogenicity) and Safety of GC3110A(Quadrivalent Influenza Vaccine)
Brief Title: A Multicenter, Double-blind, Parallel Phase III Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GC3110A_AD_P3
Record Dates: First submitted 2015-01-13; First posted 2015-02-02 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Influenza
Keywords: QIV; Quadrivalent Influenza Vaccine; Influenza vaccine; Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GC3110A(Quadrivalent) (Experimental): 0.5ml, intramuscular, a single dosing
  Interventions: Biological: GC3110A(Quadrivalent)
- GC Flu (Trivalent) (Active Comparator): 0.5ml,intramuscular,a single dosing
  Interventions: Biological: GC Flu(Trivalent)
- GC3110A(Trivalent) (Active Comparator): 0.5ml,intramuscular,a single dosing
  Interventions: Biological: GC3110A(Trivalent)

INTERVENTIONS:
Biological: GC3110A(Quadrivalent) — GC3110A(Quadrivalent), 0.5ml, intramuscular, a single dosing at Day 1
  Other Names: GC3110A
  Arms: GC3110A(Quadrivalent)
Biological: GC Flu(Trivalent) — GC Flu Pre-filled Syringe Inj.(Trivalent), 0.5ml, intramuscular, a single dosing at Day 1
  Other Names: GC Flu Pre-filled Syringe Inj.
  Arms: GC Flu (Trivalent)
Biological: GC3110A(Trivalent) — GC3110A(Trivalent), 0.5ml, intramuscular, a single dosing at Day 1
  Other Names: GC3110A
  Arms: GC3110A(Trivalent)

SUMMARY:
A Multicenter, Randomized, Double-blind, Active-controlled, Parallel Phase III

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-blind, Active-controlled, Parallel Phase III Study to Investigate the Efficacy(Immunogenicity) and Safety of GC3110A(Quadrivalent Influenza Vaccine) After Intramuscular Administration in Healthy Subjects

ELIGIBILITY:
Criteria: Inclusion Criteria:

* Given written informed consent
* Healthy Korean adults (age: over 19 )
* Korean adults who agree with 21 days follow up after vaccination and good compliance to study procedures
* Those who are able to comply with the requirements for the study

Exclusion Criteria:

* Inability in written/verbal communication
* Subjects who have participated in other interventional study within 30 days
* Alcohol or drug abuse within 6 months
* Who got the treatment of psychotropic drugs and narcotic analgesic drugs within 6 months of enrollment
* Disorders in immune function
* History of Guillain-Barré syndrome
* Disease/medications which are likely to cause any severe bleeding
* Active infection or experience of fever (>38.0 ℃) within 72 hours following vaccination
* Oral temperature >38.0 ℃ at the vaccination day
* Erythema, tattoo, injury at shoulder (vaccination site)
* Hypersensitivity with egg, chicken, or any of the vaccine components, or Neomycin, Gentamicin
* Influenza vaccination within 6months
* Any vaccination within 30 days
* Concomitant medications/therapy such as immunosuppressants or immune modifying drugs, systemic corticosteroids, immunoglobulins, blood or blood- derived products, or anti-cancer chemotherapy or radiation therapy within3 months
* Pregnant or breast-feeding women
* Clinically significant underlying diseases or medical history at investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1299 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
GMT rate of HI(Hemagglutination Inhibition) antibody for each strain | Day 21 post vaccination
  GMT (Active comparator) / GMT(Experimental)
Solicited adverse events following vaccination | Day0 up to 21 Day post vaccination
  Solicited injection site reactions: Pain, Tenderness, Erythema, Redness, Induration, and Swelling; Solicited systemic reactions: Fever, Sweating, Chill, Nausea, Vomiting, Diarrhea, Headache, Fatigue, Myalgia, Arthralgia
Unsolicited adverse events following vaccination | Day0 up to 21 Day post vaccination
  It can be estimated by Toxicity Grading Scale for healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials
SCR rate of HI(Hemagglutination Inhibition) antibody for each strain | Day 21 post vaccination
  Difference of SCR (Experimental and Active comparator)

SECONDARY OUTCOMES:
SCR rate of HI(Hemagglutination Inhibition) antibody for each strain | Day0 up to 21 Day post vaccination
SPR rate of HI(Hemagglutination Inhibition) antibody | Day 21 post vaccination
GMT rate of HI(Hemagglutination Inhibition) antibody for each strain | Day 21 post vaccination
Abnormalities in physical examination, Vital signs, clinical laboratory tests | Day 21 post vaccination
SAE | Day 180 post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Lee Jin Su, M.D, Study Director — Inha University Hospital; Choi Won Seck, M.D, Study Director — Korea University Ansan Hospital; Lee Ja Cob, Study Director — Hallym Univ. Medical Center; Woo Heong Jung, Study Director — Hallym Univ. Medical Center; Wi Sung Heon, Study Director — St Vincent's Hospital; Jeong Suk In, Study Director — Chonnam Natinal University Hospital; Kim Sin Woo, Study Director — Kyungpook National University Hospital; Kim Tae Hyung, Study Director — Soon Chun Hyang Univ. Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea